CLINICAL TRIAL: NCT04337541
Title: Reduction in COVID-19 Infection Using Surgical Facial Masks Outside the Healthcare System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Nordsjaellands Hospital (Other); Hvidovre University Hospital (Other); Herlev Hospital (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Henning Bundgaard, Professor of Cardiology, Consultant, MD, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-04-02
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The participants recruited are people working outside of their home, who have not previously been infected with COVID-19 and who do not wear facial masks (e.g. healthcare personnel) when working. They will be randomized for
  1. Normal behavior according to the authority's recommendations or
  2. Normal behavior according to the authority's recommendations and use of facial masks
  Participants will be instructed in using the facial mask consistently when outside their home (and at home when receiving visits from others. The instruction is given in writing and via an instruction video. The participants will be contacted once weekly to optimize compliance. It will be registered if the participants are diagnosed with COVID-19. Participants will perform antibody screening at study start and end. Participants, who are not tested positive for COVID-19 in the study period will perform a swab self-test if experiencing symptoms or when the study ends (instruction video).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal recommendations, no mask (No Intervention): Normal behavior according to the authority's recommendations or
- Normal recommendations AND mask (Experimental): Normal behavior according to the authority's recommendations AND use of facial masks
  Interventions: Other: Surgical facial mask

INTERVENTIONS:
Other: Surgical facial mask — Participants will follow normal Authority recommendations AND wear mask outside their homes, or when receiving visits in their home.
  Arms: Normal recommendations AND mask

SUMMARY:
In the current COVID-19 pandemic with coronavirus, SARS-COV2, the Danish Health Authorities recommend using facial masks in the health care system when handling patients presumed or proven to be infected with the virus. However, the use of facial masks outside the health care system is not recommended by the Danish Health Authorities. Here, Health Authorities in other countries have different recommendations for the use of facial masks.

Challenges when using facial masks outside the health care system include wearing the mask consistently, an efficacy of the mask of app. 8 hours necessitating a change of mask throughout the day, and that it is not sufficiently tight enough to safely keep the virus out. Moreover, the eyes (mucous membrane) remain exposed. Compliance could also be another challenge.

SARS-COV2 is assumed to primarily enter the body via the mouth through respiratory droplets - or possibly through inhalation of aerosol containing the virus. From the mouth the virus is assumed to spread to the airways and the gastro-intestinal tract. SARS-COV2 is also known to be transmitted via physical contact, helped along by the fact that the virus can survive on surfaces for at least 72 hours. Touching such a contaminated surface can transfer the virus to the mouth via the hand - and thus lead to infection of the person.

Facial masks are expected to protect against viral infection in two ways;

1. By reducing the risk of getting the virus in via the mouth or nose via respiratory droplets or aerosol
2. By reducing the transfer from virus-contaminated hands to the mouth or nose

Hypothesis The use of surgical facial masks outside the hospital will reduce the frequency of COVID-19 infection.

All participants will follow authority recommendations and be randomized to either wear facial masks or not. The participants will be screened for antibodies at study start and study end. They will perform swab-test if they experience symptoms during the study as well as the end of study.

DETAILED DESCRIPTION:
Background In the current COVID-19 pandemic with coronavirus, SARS-COV2, the Danish Health Authorities recommend using facial masks in the health care sector when handling patients presumed or proven to be infected with the virus. However, the use of facial masks outside the healthcare system is not recommended by the Danish Health Authorities. Challenges when using facial masks outside the health care system include wearing the mask consistently, an efficacy of the mask of app. 8 hours necessitating a change of mask throughout the day, and that it is not sufficiently tight enough to safely keep the virus out. Moreover, the eyes (mucous membrane) remain exposed. Compliance could also be another challenge. Health Authorities in other countries have different recommendations for the use of facial masks and the authors of the Lancet study concluded; "Universal use of face masks could be considered if supplies permit. In parallel, urgent research on the duration of protection of face masks, the measures to prolong life of disposable masks, and the invention on reusable masks should be encouraged."

SARS-COV2 is assumed to primarily enter the body via the mouth through respiratory droplets or possibly through inhalation of aerosol containing the virus. From the mouth the virus is assumed to spread to the airways and the gastro-intestinal tract. SARS-COV2 is also known to be transmitted via physical contact, helped along by the fact that the virus can survive on surfaces for at least 72 hours. Touching such a contaminated surface can transfer the virus to the mouth via the hand - and thus lead to infection of the person. A study with 26 medical students showed that they touched their face on average 23 times per hour, and that in 44 % of the incidents they touched their mucous membranes3. A Japanese questionnaire study showed that facial masks reduced the risk for school children for getting influenza by 15 %4. N95 mask and surgical facial masks are presumed to have the same effect for healthcare personnel when providing protecting from infection with influenza.

Facial masks are assumed to protect against viral infection in two ways;

1. By reducing the risk of getting the virus via mouth or nose through the air via respiratory droplets or aerosol
2. By reducing the transfer from virus-contaminated hands to the mouth or nose

About 10 % of the Danish population is estimated to get COVID-19 during the present pandemic-wave; this corresponds to 600,000 Danes. Later COVID-19 waves are expected to occur. The epidemic in Denmark is expected to be at the highest point in medio April. In April and May it be estimated that >2 % of the population will be infected per month.

Hypothesis The use of surgical facial masks outside the hospital will reduce the frequency of COVID-19 infection.

Method The participants recruited are people working outside of their home, who have not previously been infected with COVID-19 and who do not wear facial masks (e.g. healthcare personnel) when working. They will be randomized for

1. Normal behavior according to the authority's recommendations or
2. Normal behavior according to the authority's recommendations and use of facial masks

Participants will be instructed in using the facial mask consistently when outside their home (and at home when receiving visits from others. The instruction is given in writing and via an instruction video. The participants will be contacted once weekly to optimize compliance. It will be registered if the participants are diagnosed with COVID-19. Participants, who are not tested positive for COVID-19 in the study period will perform a self-test if having symptoms or when the study ends (instruction video).

Perspective The study can determine whether use of facial masks in the public is beneficial and if there is an effect this could have great impact on the current as well as any future, similar epidemics.

Interested participants can register through a link in the add to our research registration database RedCap. The participant will then receive written information and can then register. They will receive a COVID-19 screening test set and (+/-) facial masks ( 2 per day) for the first month. If the participant experience symptoms, he/she will register their symptoms in RedCap, test with a swab-test and send the swab-test to the study investigator for analyses. If negative, new test-sets are sent out - if positive, the participant will be referred to the hospital. This process continues until the participant is tested positive for COVID-19, the pandemic is considered finished by the Danish authorities or when the study ends on May 7 2020. At study end, all participants perform antibody screening and swab test, and send it to the study investigators.

Power calculation With an infection frequency of 2 % in the study period, an expected reduction of the risk to 1 % should be demonstratable with a power of 80 % and a p-value of 5 %, if including a total of 4,636 patients randomized 1:1. If the infection frequency is higher the power of the study will be higher. With an expected defection of 20 % a total of 6,000 participants will be included.

Authority approvals from The Danish National Committee On Health Research Ethics and The Data Protection Agency have been granted.

A detailed study analyses plan (SAP) will be finalized before data are analyzed.

Central registry data will be collected later when made available by national health authorities.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age and without symptoms associated with corona-virus (or previously tested positive for corona).
* Participant is outside their home more than 3 hours a day. E.g.for work or for other activities among other people.
* Do not normally wear a facial mask for daily work (e.g. healthcare personnel)

Exclusion Criteria:

* Previously tested positive for corona-virus
* Wear facial mask for work

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the difference in SARS-CoV-2 infection between the two groups after 1 months and is a combined endpoint consisting of primary outcome components 1, 2 and/or 3: | 1 month
  Component 1 of primary endpoint: Positive oropharyngeal/nasal swab with SARS-CoV-2 (PCR) and/or
The primary endpoint is the difference in SARS-CoV-2 infection between the two groups after 1 months and is a combined endpoint consisting of primary outcome components 1, 2 and/or 3: | 1 month
  Component 2 of primary endpoint: Antibody test; Development of positive SARS-CoV-2 antibody test (IgM and/or IgG) during the study period and/or
The primary endpoint is the difference in SARS-CoV-2 infection between the two groups after 1 months and is a combined endpoint consisting of primary outcome components 1, 2 and/or 3: | 1 month
  Component 3 of primary endpoint: SARS-CoV-2 infection diagnosed in a hospital/health care facility

SECONDARY OUTCOMES:
Positive oropharyngeal/nasal swab (PCR); | 1 month
  Para-influenza-virus type 1, Para-influenza-virus type 2, Human coronavirus 229E, Human coronavirus OC43, Human coronavirus NL63, Human coronavirus HKU1, Respiratory Syncytial-Virus A, Respiratory Syncytial-Virus B, Influenza A virus or Influenza B virus
Positive oropharyngeal/nasal swab (PCR); | 1 month
  SAR-CoV-2, Para-influenza-virus type 1, Para-influenza-virus type 2, Human coronavirus 229E, Human coronavirus OC43, Human coronavirus NL63, Human coronavirus HKU1, Respiratory Syncytial-Virus A, Respiratory Syncytial-Virus B, Influenza A virus or Influenza B virus

OTHER OUTCOMES:
Difference between the two study groups | 1 month
  Returned swabs
Discribtion of the face mask users psycological aspects of wearing face masks | 1 month
  Psychological aspects of face mask wearing in the community
Costs associated with wearing vs not wearing face masks | 1 month
  Cost-effectiveness analyses on the use of surgical face masks
Differences in the participants preferences | 1 month
  Preference for self-conducted home swab vs. healthcare conducted swab at hospital or similar
Difference between the two study groups | 1 month
  Symptoms of COVID-19
Difference between the two study groups with stratification between subgroups (age, gender, occupation, comorbidities) | 1 month
  Self-assessed compliance with health authority guideline on hygiene
Discribtion of the face mask users willingness to wear face masks | 1 month
  Willingness to wear face masks in the future
Healthcare diagnosed COVID-19 between study groups | 1 month
  Healthcare diagnosed COVID-19 or identified SARS-CoV-2 infection as assessed by number of participants with antibodies against SARS-CoV-2, and/or positive maso/pharyngeal swab (PCR), mortality associated with COVID-19 and all cause mortality
Hospital based diagnostics of bacteria between the two study groups | 1 month
  Presence of bacteria: Mycoplasma pneumonia, Haemophilus influenza and Legionella pneumophila (to be obtained from registries when made available)
Infection in the household between the two study groups | 1 month
  Frequency of infected house-hold members between the two groups
Sick leave among participants beteeen the two study groups | 1 month
  Frequency of sick leave between the two groups (to be obtained from registries when made available)
Predictors of primary outcome; age, gender, size of household, comorbidities, medications, social factors, occupation, mask compliance, compliance to general SARS-CoV-2 recommendations, hours outside home) | 1 month
  Predictors of primary outcome or its components

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Ullum, Prof., DMSc, Principal Investigator — Rigshospitalet, Denmark; Kasper Karmark Iversen, Prof., DMSc, Principal Investigator — Herlev Hospital; Thomas Benfield, Prof., DMSc, Principal Investigator — Hvidovre University Hospital; Christian Torp-Pedersen, Prof., DMSc, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feng S, Shen C, Xia N, Song W, Fan M, Cowling BJ. Rational use of face masks in the COVID-19 pandemic. Lancet Respir Med. 2020 May;8(5):434-436. doi: 10.1016/S2213-2600(20)30134-X. Epub 2020 Mar 20. No abstract available. PMID 32203710
- [Background] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Background] Kwok YL, Gralton J, McLaws ML. Face touching: a frequent habit that has implications for hand hygiene. Am J Infect Control. 2015 Feb;43(2):112-4. doi: 10.1016/j.ajic.2014.10.015. PMID 25637115
- [Background] Uchida M, Kaneko M, Hidaka Y, Yamamoto H, Honda T, Takeuchi S, Saito M, Kawa S. Effectiveness of vaccination and wearing masks on seasonal influenza in Matsumoto City, Japan, in the 2014/2015 season: An observational study among all elementary schoolchildren. Prev Med Rep. 2016 Dec 6;5:86-91. doi: 10.1016/j.pmedr.2016.12.002. eCollection 2017 Mar. PMID 27981021
- [Background] Gralton J, McLaws ML. Protecting healthcare workers from pandemic influenza: N95 or surgical masks? Crit Care Med. 2010 Feb;38(2):657-67. doi: 10.1097/ccm.0b013e3181b9e8b3. PMID 20095070
- [Derived] Bundgaard H, Bundgaard JS, Raaschou-Pedersen DET, von Buchwald C, Todsen T, Norsk JB, Pries-Heje MM, Vissing CR, Nielsen PB, Winslow UC, Fogh K, Hasselbalch R, Kristensen JH, Ringgaard A, Porsborg Andersen M, Goecke NB, Trebbien R, Skovgaard K, Benfield T, Ullum H, Torp-Pedersen C, Iversen K. Effectiveness of Adding a Mask Recommendation to Other Public Health Measures to Prevent SARS-CoV-2 Infection in Danish Mask Wearers : A Randomized Controlled Trial. Ann Intern Med. 2021 Mar;174(3):335-343. doi: 10.7326/M20-6817. Epub 2020 Nov 18. PMID 33205991
- [Derived] Bundgaard H, Bundgaard JS, Raaschou-Pedersen DET, Mariager AF, Schytte N, von Buchwald C, Todsen T, Skovgaard K, Trebbien R, Andersen MP, Benfield T, Ullum H, Torp-Pedersen C, Iversen K. Face masks for the prevention of COVID-19 - Rationale and design of the randomised controlled trial DANMASK-19. Dan Med J. 2020 Aug 18;67(9):A05200363. PMID 32829745